CLINICAL TRIAL: NCT02325219
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of CNTO 1959 (Guselkumab) in the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: An Efficacy and Safety of CNTO 1959 (Guselkumab) in Participants With Moderate to Severe Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103833; CNTO1959PSO3004 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; CNTO 1959; Guselkumab; Placebo
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive subcutaneous injection of CNTO 1959 50 milligram (mg) and placebo 100 mg at Week 0, 4 and then every 8 weeks thereafter.
  Interventions: Drug: CNTO 1959 50 mg; Drug: Placebo 100 mg
- Group 2 (Experimental): Participants will receive subcutaneous injection of CNTO 1959 100 milligram (mg) and placebo 50 mg at Week 0, 4 and then every 8 weeks thereafter.
  Interventions: Drug: CTNO 1959 100 mg; Drug: Placebo 50 mg
- Group 3 (Experimental): Participants will receive subcutaneous injection of placebo 50 mg and 100 mg at Weeks 0, 4 and 12. At Week 16, participants will be randomized in sub-group 3a to receive either CNTO1959 50 mg and placebo 100 mg at Week 16, 20 and then every 8 weeks thereafter or sub-group 3b to receive CNTO 1959 100 mg and placebo 50 mg at Week 16, 20 and then every 8 weeks thereafter.
  Interventions: Drug: CNTO 1959 50 mg; Drug: CTNO 1959 100 mg; Drug: Placebo 50 mg; Drug: Placebo 100 mg

INTERVENTIONS:
Drug: CNTO 1959 50 mg — Participants will receive subcutaneous injection of CNTO 1959 50 mg.
  Other Names: Guselkumab
  Arms: Group 1; Group 3
Drug: CTNO 1959 100 mg — Participants will receive subcutaneous injection of CNTO 1959 100 mg.
  Other Names: Guselkumab
  Arms: Group 2; Group 3
Drug: Placebo 50 mg — Participants will receive subcutaneous injection of Placebo matched to CNTO 1959 50 mg.
  Arms: Group 2; Group 3
Drug: Placebo 100 mg — Participants will receive subcutaneous injection of Placebo matched to CNTO 1959 100 mg.
  Arms: Group 1; Group 3

SUMMARY:
The purpose of this study is to demonstrate the superiority of CNTO 1959 (guselkumab) to placebo in the treatment of participants with moderate to severe plaque-type psoriasis (A common genetically determined, chronic, inflammatory skin disease characterized by rounded erythematous, dry, scaling patches).

DETAILED DESCRIPTION:
A Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study drug assigned by chance), double-blind (neither the Investigator nor the participant know about the study treatment), placebo-controlled (a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study of CNTO 1959 (Guselkumab) in the treatment of participants with moderate to severe plaque-type psoriasis. Participants will receive either treatment of CNTO 1959 (guselkumab) 50 milligram (mg) or 100 mg or Placebo 50 mg or 100 mg. Participants will primarily be assessed for Investigator's Global Assessment (IGA) Score and Psoriasis Area and Severity Index (PASI). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis with or without psoriatic arthritis for at least 6 months before Screening
* Have a PASI greater than or equal to (>=) 12 at Screening and at Baseline
* Have an IGA >= 3 at Screening and at Baseline
* Have an involved body surface area (BSA) >=10 percent (%) at Screening and at Baseline
* Be a candidate for phototherapy or systemic treatment for psoriasis (either naive or history of previous treatment)

Exclusion Criteria:

* Has a history of or current signs or symptoms of severe, progressive, or uncontrolled cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (example, unstable angina, atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months before Screening
* Currently has a malignancy or has a history of malignancy within 5 years before screening (with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study drug administration or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before Screening
* Has a history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance (MGUS); or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (eg, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), fungal infection (mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- Japan (27):
  - Asahikawa
  - Chūō
  - Gifu
  - Isehara
  - Izumo
  - Kanazawa
  - Kawasaki
  - Kita-Gun
  - Kochi
  - Kurume
  - Kyoto
  - Matsumoto
  - Miyagi
  - Morioka
  - Nagoya
  - Osaka
  - Ōsaka-sayama
  - Sapporo
  - Shimotsuke
  - Shinjuku-ku
  - Tokushima
  - Tokyo
  - Tōon
  - Tsu
  - Tsukuba
  - Ube
  - Yokosuka

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Controlled Period [CP]): Participants stratified by the type of psoriasis (with or without PsA) received placebo 50 milligram (mg) and 100 mg as subcutaneous (SC) injection at Week 0, Week 4, and Week 12. At Week 16, participants in the placebo group were re-randomized to receive either guselkumab 50 mg or guselkumab 100 mg, stratified by the type of psoriasis (with or without psoriatic arthritis [PsA]).
- Guselkumab 50 mg (CP): Participants stratified by the type of psoriasis (with or without PsA) received guselkumab 50 mg SC injection and placebo 100 mg at Week 0, Week 4, and Week 12. Participants who completed CP continued to after CP period. At Week 16, participants in this group received placebo 50 mg and 100 mg to maintain blind. After Week 16, participants received guselkumab 50 mg and placebo 100 mg at Weeks 20, 28, 36, and 44 after CP.
- Guselkumab 100 mg (CP): Participants stratified by the type of psoriasis (with or without PsA) received guselkumab 100 mg SC injection and placebo 50 mg at Week 0, Week 4, and Week 12. Participants who completed CP continued to after CP period. At Week 16, participants in this group received placebo 50 mg and 100 mg to maintain blind. After Week 16, participants received guselkumab 100 mg and placebo 50 mg at Weeks 20, 28, 36, and 44 after CP.
- Placebo to Guselkumab 50 mg (After CP): Participants (who received placebo in CP and re-randomized at Week 16) received guselkumab 50 mg and placebo 100 mg at Weeks 16, 20, 28, 36, and 44.
- Placebo to Guselkumab 100 mg (After CP): Participants (who received placebo in CP and re-randomized at Week 16) received guselkumab 100 mg and placebo 50 mg at Weeks 16 20, 28, 36, and 44.
Period: Controlled Period (Week 0 - 16)
Arm/Group | Placebo (Controlled Period [CP]) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Started | 64 | 65 | 63 | 0 | 0
Completed | 52 | 63 | 62 | 0 | 0
Not Completed | 12 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 6 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: After Controlled Period (Week 16 - 52)
Arm/Group | Placebo (Controlled Period [CP]) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Started | 0 | 63 | 62 | 26 (Participants who completed CP and re-randomized to Guselkumab 50 mg.) | 26 (Participants who completed CP and re-randomized to Guselkumab 100 mg.)
Completed | 0 | 60 | 62 | 26 | 25
Not Completed | 0 | 3 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (CP): Participants received placebo 50 milligram (mg) and 100 mg as subcutaneous (SC) injection at Week 0, Week 4, and Week 12. At Week 16, participants in the placebo group were re-randomized to receive either guselkumab 50 mg or guselkumab 100 mg, stratified by the type of psoriasis (with or without psoriatic arthritis [PsA]).
- Total: Total of all reporting groups
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Total
Number analyzed (Participants) | 64 | 65 | 63 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (10.56) | 50.1 (12.66) | 47.8 (11.07) | 48.8 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 16 | 47
  Male | 54 | 44 | 47 | 145
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 64 | 65 | 63 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16
Description: The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 16
Population: The randomized analysis set included all randomized participants at Week 0, regardless of whether or not they received the study treatment and had any postbaseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants | 7.8 | 92.3 | 88.9
Statistical Analysis 1: Comparison: Placebo (CP) vs Guselkumab 50 mg (CP); Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo (CP) vs Guselkumab 100 mg (CP); Test type: Superiority; p < 0.001, Fisher Exact

2. Primary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI) 90 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 90 response was defined as at least a 90% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants | 0 | 70.8 | 69.8
Statistical Analysis 1: Comparison: Placebo (CP) vs Guselkumab 50 mg (CP); Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo (CP) vs Guselkumab 100 mg (CP); Test type: Superiority; p < 0.001, Fisher Exact

3. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 75 response was defined as at least a 75% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants | 6.3 | 89.2 | 84.1

4. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale | -0.8 (5.40) | -8.3 (5.87) | -8.5 (6.95)

5. Secondary Outcome: Percentage of Participants With an IGA Score of Cleared (0), Cleared (0) or Minimal (1), and Cleared (0) or Minimal (1) or Mild (2) at Weeks 2, 4, 8, 12, and 16
Description: as for outcome 1
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants
  Week 2: IGA 0 responders | 0 | 0 | 0
  Week 2: IGA 0/1 responders | 0 | 3.1 | 9.5
  Week 2: IGA 0/1/2 responders | 10.9 | 47.7 | 46.0
  Week 4: IGA 0 responders | 0 | 1.5 | 6.3
  Week 4: IGA 0/1 responders | 1.6 | 27.7 | 25.4
  Week 4: IGA 0/1/2 responders | 20.3 | 81.5 | 77.8
  Week 8: IGA 0 responders | 0 | 16.9 | 20.6
  Week 8: IGA 0/1 responders | 1.6 | 76.9 | 65.1
  Week 8: IGA 0/1/2 responders | 20.3 | 93.8 | 93.7
  Week 12: IGA 0 responders | 0 | 33.8 | 33.3
  Week 12: IGA 0/1 responders | 4.7 | 89.2 | 84.1
  Week 12: IGA 0/1/2 responders | 25.0 | 95.4 | 96.8
  Week 16: IGA 0 responders | 0 | 44.6 | 44.4
  Week 16: IGA 0/1 responders | 7.8 | 92.3 | 88.9
  Week 16: IGA 0/1/2 responders | 28.1 | 96.9 | 96.8

6. Secondary Outcome: Percentage of Participants With an IGA Score of Cleared (0), Cleared (0) or Minimal (1), and Cleared (0) or Minimal (1) or Mild (2) at Weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52
Description: as for outcome 1
Time Frame: Weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: The analysis population for this time frame included all participants who were randomized to Guselkumab at Week 0 or 16, regardless of whether or not they received the study treatment and had any postbaseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
percentage of participants
  Week 20: IGA 0 responders | 46.2 | 57.1 | 3.8 | 11.5
  Week 20: IGA 0/1 responders | 89.2 | 92.1 | 57.7 | 46.2
  Week 20: IGA 0/1/2 responders | 96.9 | 96.8 | 84.6 | 88.5
  Week 24: IGA 0 responders | 53.8 | 57.1 | 15.4 | 38.5
  Week 24: IGA 0/1 responders | 90.8 | 88.9 | 88.5 | 80.8
  Week 24: IGA 0/1/2 responders | 98.5 | 96.8 | 96.2 | 100.0
  Week 28: IGA 0 responders | 53.8 | 49.2 | 50.0 | 46.2
  Week 28: IGA 0/1 responders | 90.8 | 88.9 | 100.0 | 88.5
  Week 28: IGA 0/1/2 responders | 98.5 | 95.2 | 100.0 | 100.0
  Week 32: IGA 0 responders | 47.7 | 55.6 | 53.8 | 50.0
  Week 32: IGA 0/1 responders | 89.2 | 90.5 | 100.0 | 92.3
  Week 32: IGA 0/1/2 responders | 98.5 | 96.8 | 100.0 | 100.0
  Week 36: IGA 0 responders | 44.6 | 55.6 | 61.5 | 46.2
  Week 36: IGA 0/1 responders | 89.2 | 90.5 | 100.0 | 92.3
  Week 36: IGA 0/1/2 responders | 98.5 | 96.8 | 100.0 | 100.0
  Week 40: IGA 0 responders | 49.2 | 55.6 | 65.4 | 57.7
  Week 40: IGA 0/1 responders | 87.7 | 92.1 | 100.0 | 92.3
  Week 40: IGA 0/1/2 responders | 96.9 | 98.4 | 100.0 | 100.0
  Week 44: IGA 0 responders | 55.4 | 52.4 | 61.5 | 57.7
  Week 44: IGA 0/1 responders | 86.2 | 88.9 | 100.0 | 92.3
  Week 44: IGA 0/1/2 responders | 98.5 | 96.8 | 100.0 | 100.0
  Week 48: IGA 0 responders | 50.8 | 60.3 | 73.1 | 57.7
  Week 48: IGA 0/1 responders | 86.2 | 87.3 | 100.0 | 92.3
  Week 48: IGA 0/1/2 responders | 98.5 | 96.8 | 100.0 | 100.0
  Week 52: IGA 0 responders | 53.8 | 58.7 | 53.8 | 50.0
  Week 52: IGA 0/1 responders | 87.7 | 90.5 | 100.0 | 88.5
  Week 52: IGA 0/1/2 responders | 98.5 | 98.4 | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants Who Achieved PASI 50, PASI 75, PASI 90, and PASI 100 Responses at Weeks 2, 4, 8, 12, and 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 50, 75, 90, and 100 responses were defined as at least a 50%, 75%, 90%, and 100% reduction in PASI relative to Baseline respectively.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants
  Week 2: PASI 50 responders | 0 | 4.6 | 17.5
  Week 2: PASI 75 responders | 0 | 0 | 1.6
  Week 2: PASI 90 responders | 0 | 0 | 0
  Week 2: PASI 100 responders | 0 | 0 | 0
  Week 4: PASI 50 responders | 1.6 | 49.2 | 49.2
  Week 4: PASI 75 responders | 0 | 15.4 | 17.5
  Week 4: PASI 90 responders | 0 | 4.6 | 4.8
  Week 4: PASI 100 responders | 0 | 1.5 | 1.6
  Week 8: PASI 50 responders | 9.4 | 87.7 | 79.4
  Week 8: PASI 75 responders | 0 | 55.4 | 50.8
  Week 8: PASI 90 responders | 0 | 30.8 | 30.2
  Week 8: PASI 100 responders | 0 | 7.7 | 7.9
  Week 12: PASI 50 responders | 7.8 | 90.8 | 92.1
  Week 12: PASI 75 responders | 3.1 | 78.5 | 79.4
  Week 12: PASI 90 responders | 0 | 47.7 | 38.1
  Week 12: PASI 100 responders | 0 | 16.9 | 22.2
  Week 16: PASI 50 responders | 14.1 | 93.8 | 95.2
  Week 16: PASI 75 responders | 6.3 | 89.2 | 84.1
  Week 16: PASI 90 responders | 0 | 70.8 | 69.8
  Week 16: PASI 100 responders | 0 | 32.3 | 27.0

8. Secondary Outcome: Percentage of Participants Who Achieved PASI 50, PASI 75, PASI 90, and PASI 100 Responses at Weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52
Description: as for outcome 7
Time Frame: Weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
percentage of participants
  Week 20: PASI 50 responders | 95.4 | 96.8 | 57.7 | 65.4
  Week 20: PASI 75 responders | 90.8 | 88.9 | 46.2 | 30.8
  Week 20: PASI 90 responders | 70.8 | 71.4 | 19.2 | 15.4
  Week 20: PASI 100 responders | 33.8 | 34.9 | 3.8 | 0
  Week 24: PASI 50 responders | 98.5 | 98.4 | 92.3 | 84.6
  Week 24: PASI 75 responders | 90.8 | 90.5 | 80.8 | 61.5
  Week 24: PASI 90 responders | 78.5 | 76.2 | 42.3 | 46.2
  Week 24: PASI 100 responders | 41.5 | 44.4 | 11.5 | 23.1
  Week 28: PASI 50 responders | 98.5 | 98.4 | 100.0 | 92.3
  Week 28: PASI 75 responders | 92.3 | 90.5 | 88.5 | 80.8
  Week 28: PASI 90 responders | 75.4 | 77.8 | 73.1 | 61.5
  Week 28: PASI 100 responders | 44.6 | 38.1 | 30.8 | 34.6
  Week 32: PASI 50 responders | 98.5 | 98.4 | 100.0 | 96.2
  Week 32: PASI 75 responders | 92.3 | 90.5 | 92.3 | 84.6
  Week 32: PASI 90 responders | 76.9 | 76.2 | 76.9 | 69.2
  Week 32: PASI 100 responders | 41.5 | 44.4 | 34.6 | 38.5
  Week 36: PASI 50 responders | 98.5 | 95.2 | 100.0 | 96.2
  Week 36: PASI 75 responders | 92.3 | 90.5 | 96.2 | 92.3
  Week 36: PASI 90 responders | 78.5 | 76.2 | 84.6 | 65.4
  Week 36: PASI 100 responders | 36.9 | 42.9 | 30.8 | 42.3
  Week 40: PASI 50 responders | 98.5 | 98.4 | 100.0 | 96.2
  Week 40: PASI 75 responders | 90.8 | 90.5 | 100.0 | 92.3
  Week 40: PASI 90 responders | 78.5 | 77.8 | 96.2 | 73.1
  Week 40: PASI 100 responders | 33.8 | 44.4 | 38.5 | 50.0
  Week 44: PASI 50 responders | 98.5 | 95.2 | 100.0 | 96.2
  Week 44: PASI 75 responders | 90.8 | 88.9 | 100.0 | 92.3
  Week 44: PASI 90 responders | 80.0 | 74.6 | 88.5 | 73.1
  Week 44: PASI 100 responders | 38.5 | 44.4 | 42.3 | 50.0
  Week 48: PASI 50 responders | 98.5 | 96.8 | 100.0 | 96.2
  Week 48: PASI 75 responders | 90.8 | 93.7 | 100.0 | 92.3
  Week 48: PASI 90 responders | 75.4 | 77.8 | 100.0 | 76.9
  Week 48: PASI 100 responders | 36.9 | 49.2 | 46.2 | 42.3
  Week 52: PASI 50 responders | 98.5 | 98.4 | 100.0 | 96.2
  Week 52: PASI 75 responders | 92.3 | 90.5 | 100.0 | 92.3
  Week 52: PASI 90 responders | 75.4 | 77.8 | 92.3 | 73.1
  Week 52: PASI 100 responders | 38.5 | 47.6 | 38.5 | 42.3

9. Secondary Outcome: Percent Change From Baseline in the PASI Total Score at Weeks 2, 4, 8, 12, 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percent change
  Week 2 | 0.4 (18.55) | 20.1 (20.85) | 23.6 (23.76)
  Week 4 | 0.0 (27.74) | 45.3 (26.72) | 44.9 (30.80)
  Week 8 | 1.5 (32.73) | 74.5 (22.39) | 70.3 (25.42)
  Week 12 | 0.5 (38.28) | 83.7 (20.00) | 82.9 (18.56)
  Week 16 | 0.2 (45.53) | 88.9 (17.34) | 88.7 (17.77)

10. Secondary Outcome: Percent Change From Baseline in the PASI Total Score at Weeks 20, 24, 28, 22, 36, 40, 44, 48, and 52
Description: as for outcome 9
Time Frame: Baseline and Weeks 20, 24, 28, 22, 36, 40, 44, 48, and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
percent change
  Week 20 | 89.4 (18.21) | 90.6 (16.45) | 58.7 (33.67) | 51.9 (39.06)
  Week 24 | 91.6 (14.59) | 92.1 (15.51) | 80.7 (24.87) | 78.8 (22.44)
  Week 28 | 91.9 (14.05) | 91.4 (16.24) | 91.6 (10.81) | 85.6 (20.60)
  Week 32 | 92.5 (12.38) | 92.0 (15.78) | 93.1 (8.59) | 89.1 (19.66)
  Week 36 | 92.2 (13.42) | 90.5 (19.40) | 94.7 (6.76) | 91.5 (13.84)
  Week 40 | 92.3 (13.86) | 92.1 (15.86) | 96.4 (3.87) | 92.3 (14.08)
  Week 44 | 91.8 (17.30) | 91.1 (17.26) | 96.6 (4.39) | 92.2 (14.28)
  Week 48 | 91.5 (17.28) | 92.1 (16.14) | 97.9 (2.73) | 91.8 (14.21)
  Week 52 | 91.6 (17.12) | 92.5 (15.39) | 96.7 (4.45) | 91.4 (14.02)

11. Secondary Outcome: Change From Baseline in the PASI Total Score at Weeks 2, 4, 8, 12, 16
Description: as for outcome 9
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale
  Week 2 | 0.0 (4.44) | -5.7 (7.13) | -6.3 (7.17)
  Week 4 | -0.2 (7.13) | -12.1 (10.55) | -12.5 (11.00)
  Week 8 | -1.0 (8.99) | -19.1 (10.62) | -19.2 (11.80)
  Week 12 | -0.6 (10.62) | -21.4 (11.11) | -22.4 (11.86)
  Week 16 | -0.5 (12.39) | -22.6 (11.00) | -23.9 (12.27)

12. Secondary Outcome: Change From Baseline in the PASI Total Score at Weeks 20, 24, 28, 32, 36, 40, 44, 48, 52
Description: as for outcome 9
Time Frame: Baseline and Weeks 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 20 | -22.8 (11.23) | -24.3 (12.52) | -18.3 (15.46) | -11.3 (10.33)
  Week 24 | -23.4 (11.16) | -24.7 (12.35) | -24.2 (15.12) | -18.2 (9.56)
  Week 28 | -23.6 (11.44) | -24.5 (12.56) | -27.0 (14.84) | -20.1 (10.52)
  Week 32 | -23.7 (11.30) | -24.7 (12.58) | -27.6 (15.02) | -21.0 (11.05)
  Week 36 | -23.6 (11.38) | -24.3 (12.72) | -28.0 (15.02) | -21.5 (10.37)
  Week 40 | -23.7 (11.51) | -24.6 (12.29) | -28.4 (14.96) | -21.7 (10.65)
  Week 44 | -23.5 (11.69) | -24.3 (12.29) | -28.5 (15.04) | -21.6 (10.55)
  Week 48 | -23.4 (11.59) | -24.6 (12.27) | -28.7 (14.90) | -21.6 (10.78)
  Week 52 | -23.5 (11.74) | -24.6 (12.11) | -28.5 (15.07) | -21.5 (10.62)

13. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Involvement by Psoriatic Lesions at Week 48
Description: BSA as physical measure to define disease severity is to determine how much of the Body Surface Area (BSA) is affected by psoriasis. Involved BSA is calculated by using the palm of the participant's hand as equivalent to 1% of the BSA (rule of palm). Psoriasis affected BSA under 5% suggests mild psoriasis, a BSA of 5% to 10% is considered moderate, and an involved BSA of over 10% indicates severe psoriasis.
Time Frame: Baseline and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Change in BSA (% points)
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
Change in BSA (% points) | -31.7 (22.40) | -34.4 (21.19) | -37.1 (22.24) | -27.7 (16.08)

14. Secondary Outcome: Change From Baseline in Nail Psoriasis Area and Severity Index (NAPSI) Score at Week 16
Description: NAPSI is an index used for assessing and grading the severity of nail psoriasis. A target nail representing the worst nail psoriasis at baseline is divided into quadrants and is graded for nail matrix psoriasis (pitting, leukonychia, red spots in the lunula, and nail plate crumbling) and nail bed psoriasis (onycholysis, splinter hemorrhages, oil drop discoloration, and nail bed hyperkeratosis), each on a scale of 0 to 4. The sum of these scores is the total NAPSI score. The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 (no psoriasis) to 80 (psoriasis present in all 4 quadrants of all 10 nails).
Time Frame: Baseline and Week 16
Population: Population included participants randomized at Week 0 and with nail psoriasis at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 42 | 44 | 40
units on a scale | -0.2 (1.13) | -1.2 (1.61) | -1.5 (1.78)

15. Secondary Outcome: Change From Baseline in NAPSI Score at Weeks 28, 36, 48, 52
Description: as for outcome 14
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: Population included participants randomized to Guselkumab at Week 0 or 16 and with nail psoriasis at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 44 | 40 | 15 | 18
units on a scale
  Week 28 | -2.2 (1.79) | -2.4 (2.34) | -1.7 (1.40) | -0.7 (1.13)
  Week 36 | -2.3 (2.01) | -2.7 (2.23) | -2.5 (1.77) | -1.2 (1.50)
  Week 48 | -2.7 (1.91) | -2.7 (2.44) | -3.3 (2.22) | -1.7 (1.75)
  Week 52 | -2.8 (1.94) | -2.7 (2.20) | -3.3 (2.34) | -1.4 (1.54)

16. Secondary Outcome: Percent Change From Baseline in NAPSI Score at Week 16
Description: as for outcome 14
Time Frame: Baseline and Week 16
Population: Population included participants randomized at Week 0 and with nail psoriasis at baseline.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 42 | 44 | 40
percent change | 1.0 (59.38) | 31.6 (43.56) | 39.1 (48.93)

17. Secondary Outcome: Percent Change From Baseline in NAPSI Score at Weeks 28, 36, 48, 52
Description: as for outcome 14
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: Population included participants randomized to Guselkumab at Week 0 or 16 and with nail psoriasis at baseline.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 44 | 40 | 15 | 18
percent change
  Week 28 | 57.9 (42.99) | 61.1 (43.15) | 48.7 (38.77) | 23.6 (49.69)
  Week 36 | 59.6 (46.95) | 67.4 (45.44) | 69.9 (30.48) | 38.4 (40.34)
  Week 48 | 71.0 (37.11) | 68.1 (49.01) | 80.2 (23.06) | 53.7 (42.99)
  Week 52 | 74.4 (35.11) | 75.3 (41.32) | 79.2 (25.62) | 44.9 (53.56)

18. Secondary Outcome: Percentage of Participants With a Scalp-specific Investigator's Global Assessment (Ss-IGA) Score of 0 or 1 and at Least a 2-grade Improvement From Baseline at Week 16
Description: The percentage of participants with an ss-IGA score of absence of disease (0) or very mild disease (1) and at least a 2-grade improvement from Baseline at Week 16 among participants who had an ss-IGA score of >= 2 at baseline was evaluated. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: Absence of Disease (0), Very Mild Disease (1), Mild Disease (2), Moderate Disease (3), and Severe Disease (4).
Time Frame: Week 16
Population: Population included participants randomized at Week 0 and with baseline ss-IGA score >= 2.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 57 | 58 | 58
percentage of participants | 10.5 | 74.1 | 82.8

19. Secondary Outcome: Percentage of Participants With an Ss-IGA Score of 0 or 1 and at Least a 2-grade Improvement From Baseline at Weeks 28, 48 and 52
Description: as for outcome 18
Time Frame: Week 28, 48 and 52
Population: Population included participants randomized to Guselkumab at Week 0 or 16 and with baseline ss-IGA score >= 2.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 58 | 58 | 21 | 24
percentage of participants
  Week 28 | 86.2 | 86.2 | 90.5 | 70.8
  Week 48 | 84.5 | 84.5 | 85.7 | 83.3
  Week 52 | 84.5 | 86.2 | 85.7 | 95.8

20. Secondary Outcome: Percentage of Participants Who Achieved Ss-IGA Scores Among Participants With Baseline Ss-IGA Score >=2 at Week 16
Description: The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: Absence of Disease (0), Very Mild Disease (1), Mild Disease (2), Moderate Disease (3), and Severe Disease (4).
Time Frame: Week 16
Population: Population included participants randomized at Week 0 and with baseline ss-IGA score >= 2.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 57 | 58 | 58
percentage of participants
  Absence of Disease (0) | 3.5 | 48.3 | 63.8
  Very Mild Disease (1) | 8.8 | 41.4 | 22.4
  Mild Disease (2) | 21.1 | 8.6 | 8.6
  Moderate Disease (3) | 49.1 | 1.7 | 5.2
  Severe Disease (4) | 17.5 | 0 | 0

21. Secondary Outcome: Percentage of Participants Who Achieved Ss-IGA Scores Among Participants With Baseline Ss-IGA Score >=2 at Week 28, 48 and 52
Description: as for outcome 20
Time Frame: Week 28, 48 and 52
Population: Population included participants randomized to Guselkumab at Week 0 or 16 and with baseline ss-IGA score >= 2
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 58 | 58 | 21 | 24
percentage of participants
  Week 28: Absence of Disease (0) | 63.8 | 70.7 | 66.7 | 50.0
  Week 28: Very Mild Disease (1) | 31.0 | 22.4 | 28.6 | 25.0
  Week 28: Mild Disease (2) | 3.4 | 3.4 | 4.8 | 12.5
  Week 28: Moderate Disease (3) | 1.7 | 3.4 | 0 | 12.5
  Week 28: Severe Disease (4) | 0 | 0 | 0 | 0
  Week 48: Absence of Disease (0) | 67.2 | 75.9 | 76.2 | 66.7
  Week 48: Very Mild Disease (1) | 25.9 | 13.8 | 9.5 | 20.8
  Week 48: Mild Disease (2) | 5.2 | 6.9 | 9.5 | 12.5
  Week 48: Moderate Disease (3) | 1.7 | 3.4 | 4.8 | 0
  Week 48: Severe Disease (4) | 0 | 0 | 0 | 0
  Week 52: Absence of Disease (0) | 67.2 | 77.6 | 66.7 | 75.0
  Week 52: Very Mild Disease (1) | 27.6 | 10.3 | 19.0 | 20.8
  Week 52: Mild Disease (2) | 3.4 | 10.3 | 14.3 | 4.2
  Week 52: Moderate Disease (3) | 1.7 | 1.7 | 0 | 0
  Week 52: Severe Disease (4) | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Weeks 8 and 16
Description: as for outcome 4
Time Frame: Weeks 8 and 16
Population: Population included participants randomized at Week 0 and with baseline DLQI > 1.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 61 | 64 | 60
percentage of participants
  Week 8 | 6.6 | 43.8 | 43.3
  Week 16 | 6.6 | 64.1 | 68.3

23. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Weeks 28, 36, 48, and 52
Description: as for outcome 4
Time Frame: Weeks 28, 36, 48, and 52
Population: Population included participants randomized to Guselkumab at Week 0 or 16 and with baseline DLQI <=1.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 64 | 60 | 24 | 25
percentage of participants
  Week 28 | 70.3 | 75.0 | 50.0 | 68.0
  Week 36 | 79.7 | 83.3 | 79.2 | 68.0
  Week 48 | 73.4 | 73.3 | 62.5 | 72.0
  Week 52 | 73.4 | 76.7 | 75.0 | 80.0

24. Secondary Outcome: Change From Baseline in the DLQI Total Score at Week 8
Description: as for outcome 4
Time Frame: Baseline and Weeks 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale | -0.4 (4.71) | -7.5 (5.28) | -7.0 (6.35)

25. Secondary Outcome: Change From Baseline in the DLQI Total Score at Weeks 28, 36, 48, 52
Description: as for outcome 4
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 28 | -9.0 (5.85) | -8.9 (6.95) | -9.5 (7.73) | -5.5 (5.19)
  Week 36 | -9.2 (6.44) | -9.2 (7.27) | -10.3 (8.01) | -6.1 (5.99)
  Week 48 | -9.2 (6.20) | -9.1 (7.12) | -10.1 (7.94) | -6.1 (5.82)
  Week 52 | -9.2 (6.39) | -9.0 (7.28) | -10.1 (7.79) | -6.5 (5.05)

26. Secondary Outcome: Percentage of Participants With >=5-point Decrease in the DLQI Total Score From Baseline at Weeks 8 and 16
Description: as for outcome 4
Time Frame: Weeks 8 and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
percentage of participants
  Week 8 | 17.2 | 61.5 | 58.7
  Week 16 | 20.3 | 67.7 | 69.8

27. Secondary Outcome: Percentage of Participants With >=5-point Decrease in the DLQI Total Score From Baseline at Weeks 28, 36, 48, and 52
Description: as for outcome 4
Time Frame: Weeks 28, 36, 48, and 52
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
percentage of participants
  Week 28 | 69.2 | 73.0 | 65.4 | 57.7
  Week 36 | 72.3 | 68.3 | 69.2 | 57.7
  Week 48 | 72.3 | 71.4 | 69.2 | 61.5
  Week 52 | 72.3 | 71.4 | 69.2 | 61.5

28. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions Questionnaire (EQ-5D): Index Score at Week 16
Description: The EQ-5D is designed for self-completion by participants and consists of 2 pages - the EQ-5D descriptive system and the EQ visual analog scale (EQ VAS). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and severe problems. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale | 0.05 (0.141) | 0.20 (0.199) | 0.18 (0.210)

29. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions Questionnaire (EQ-5D): Index Score at Weeks 28 and 48
Description: as for outcome 28
Time Frame: Baseline and Weeks 28, 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 28 | 0.20 (0.187) | 0.20 (0.221) | 0.25 (0.170) | 0.14 (0.133)
  Week 48 | 0.20 (0.198) | 0.21 (0.228) | 0.28 (0.152) | 0.15 (0.140)

30. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) at Week 16
Description: The EQ visual analog scale (EQ VAS) is the part of EQ-5D scale. The EQ VAS records the respondent's self-rated health on a vertical, visual analog scale where the endpoints are labeled 'Best imaginable health state' (score of 100) and 'Worst imaginable health state' (score of 0).
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale | 2.45 (22.440) | 21.20 (23.542) | 18.43 (26.206)

31. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) at Weeks 28, 48
Description: as for outcome 30
Time Frame: Baseline and Weeks 28, 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 28 | 22.94 (24.759) | 20.87 (26.465) | 20.73 (20.095) | 11.62 (26.831)
  Week 48 | 20.88 (29.647) | 21.70 (26.577) | 20.38 (22.094) | 7.00 (29.490)

32. Secondary Outcome: Change From Baseline in the Physical and Mental Component Summary (PCS and MCS) Scores of 36- Item Short Form Health Assessment Questionnaire (SF-36) at Week 16
Description: SF-36 V2 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. Higher scores indicate better health status.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale
  PCS | 0.3 (9.90) | 7.4 (15.65) | 7.3 (14.40)
  MCS | 1.3 (8.21) | 4.0 (7.22) | 5.3 (9.63)

33. Secondary Outcome: Change From Baseline in the PCS and MCS Scores of 36- Item Short Form Health Assessment Questionnaire (SF-36) at Weeks 28 and 48
Description: SF-36 V2 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: PCS and MCS. The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. Higher scores indicate better health status.
Time Frame: Baseline and Weeks 28, 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 28: PCS | 7.7 (13.71) | 8.9 (14.83) | 6.4 (10.20) | 5.4 (9.80)
  Week 48: PCS | 8.2 (14.22) | 8.4 (15.16) | 8.8 (12.13) | 4.4 (7.60)
  Week 28: MCS | 5.9 (9.62) | 4.6 (10.30) | 6.5 (6.91) | 4.9 (9.83)
  Week 48: MCS | 5.7 (9.04) | 5.6 (9.32) | 4.5 (9.92) | 5.0 (11.00)

34. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire Scores at Week 16
Description: Changes from baseline in the 4 types (absenteeism, activity impairment, presenteeism, and Work productivity loss) of WPAI scores at Week 16 were evaluated. The WPAI questionnaire is used to measure productivity loss associated with psoriasis during the past 7 days. It consists of six questions about absence from work because of psoriasis, hours actually worked, reduction in productivity at work attributed to psoriasis and reduction in productivity while performing daily activities. Four separate overall scores were calculated, including absenteeism (work time missed due to health), presenteeism (impairment at work due to health), work productivity loss (overall work impairment due to health), and activity impairment due to health. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity.
Time Frame: Baseline and Week 16
Population: The randomized analysis set included all randomized participants at Week 0, regardless of whether or not they received the study treatment and had any postbaseline efficacy assessment. Here 'n' (number analyzed) signifies the number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 64 | 65 | 63
units on a scale
  Absenteeism: number analyzed (Participants) | 58 | 55 | 51
  Absenteeism | 0.9 (14.96) | -2.4 (8.14) | -1.9 (8.18)
  Activity Impairment | -7.7 (24.09) | -30.9 (31.95) | -33.8 (33.91)
  Presenteeism: number analyzed (Participants) | 58 | 54 | 51
  Presenteeism | -7.2 (22.62) | -22.0 (34.06) | -23.7 (30.92)
  Work Productivity Loss: number analyzed (Participants) | 58 | 54 | 51
  Work Productivity Loss | -7.6 (23.24) | -23.0 (34.38) | -24.1 (31.79)

35. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire Scores at Weeks 28 and 48
Description: Changes from baseline in the 4 types (absenteeism, activity impairment, presenteeism, and Work productivity loss) of WPAI scores at Weeks 28 and 48 were evaluated. The WPAI questionnaire is used to measure productivity loss associated with psoriasis during the past 7 days. It consists of six questions about absence from work because of psoriasis, hours actually worked, reduction in productivity at work attributed to psoriasis and reduction in productivity while performing daily activities. Four separate overall scores were calculated, including absenteeism (work time missed due to health), presenteeism (impairment at work due to health), work productivity loss (overall work impairment due to health), and activity impairment due to health. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity.
Time Frame: Baseline and Weeks 28, 48
Population: The analysis population for this time frame included all participants who were randomized to Guselkumab at Week 0 or 16, regardless of whether or not they received the study treatment and had any postbaseline efficacy assessment. Here 'n' signifies the number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 65 | 63 | 26 | 26
units on a scale
  Week 28: Absenteeism: number analyzed (Participants) | 55 | 51 | 24 | 23
  Week 28: Absenteeism | -3.0 (10.93) | -2.8 (9.12) | -4.0 (8.78) | -0.1 (2.03)
  Week 28: Activity Impairment | -35.1 (32.02) | -33.5 (32.19) | -32.7 (29.20) | -28.1 (28.85)
  Week 28: Presenteeism: number analyzed (Participants) | 54 | 51 | 24 | 23
  Week 28: Presenteeism | -26.9 (30.83) | -24.5 (34.43) | -27.1 (25.62) | -18.7 (26.85)
  Week 28: Work Productivity Loss: number analyzed (Participants) | 54 | 51 | 24 | 23
  Week 28: Work Productivity Loss | -28.1 (31.18) | -25.1 (35.05) | -28.3 (26.61) | -18.3 (26.68)
  Week 48: Absenteeism: number analyzed (Participants) | 55 | 51 | 24 | 23
  Week 48: Absenteeism | -2.0 (6.56) | -2.9 (9.37) | -4.5 (9.02) | 0.7 (2.49)
  Week 48: Activity Impairment | -38.0 (30.58) | -36.8 (31.72) | -36.2 (28.44) | -25.0 (30.50)
  Week 48: Presenteeism: number analyzed (Participants) | 54 | 51 | 24 | 23
  Week 48: Presenteeism | -29.3 (31.25) | -30.8 (30.97) | -30.0 (29.93) | -20.4 (27.88)
  Week 48: Work Productivity Loss: number analyzed (Participants) | 54 | 51 | 24 | 23
  Week 48: Work Productivity Loss | -29.6 (31.88) | -31.4 (31.71) | -31.5 (30.93) | -19.2 (27.84)

36. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 20, ACR 50, and ACR 70 Responses at Weeks 4, 8, and 16
Description: ACR Response is defined as percent improvement from baseline of 20%, 50%, and 70% (ACR20, ACR50, and ACR70, respectively) in swollen joint (66 joints) and tender joint (68 joints) counts and percent improvement from baseline of 20%, 50%, and 70% (ACR20, ACR50, and ACR70, respectively) in 3 of following 5 assessments: patient's assessment of pain using VAS (VAS; 0-10, 0=no pain and 10=worst possible pain), patient's global assessment of disease activity by using VAS (scale ranges from 0 to 10, 0=very well and 10=very poor), physician's global assessment of disease activity using VAS (0=no arthritis activity and 10 = extremely active arthritis), patient's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Weeks 4, 8, and 16
Population: Population included randomized participants at Week 0 and who had a diagnosis of PsA at screening.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 10
percentage of participants
  Week 4: ACR 20 responders | 0 | 27.3 | 10.0
  Week 4: ACR 50 responders | 0 | 18.2 | 0
  Week 4: ACR 70 responders | 0 | 9.1 | 0
  Week 8: ACR 20 responders | 10.0 | 45.5 | 20.0
  Week 8: ACR 50 responders | 0 | 36.4 | 20.0
  Week 8: ACR 70 responders | 0 | 18.2 | 0
  Week 16: ACR 20 responders | 0 | 45.5 | 30.0
  Week 16: ACR 50 responders | 0 | 18.2 | 30.0
  Week 16: ACR 70 responders | 0 | 9.1 | 30.0

37. Secondary Outcome: Percentage of Participants Who Achieved ACR 20, ACR 50, and ACR 70 Responses at Weeks 28, 36, 48, and 52
Description: as for outcome 36
Time Frame: Weeks 28, 36, 48, and 52
Population: Population included participants who were randomized to Guselkumab at Week 0 or 16 and had a diagnosis of PsA at screening.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 10 | 3 | 4
percentage of participants
  Week 28: ACR 20 responders | 36.4 | 40.0 | 66.7 | 0
  Week 28: ACR 50 responders | 27.3 | 40.0 | 33.3 | 0
  Week 28: ACR 70 responders | 18.2 | 30.0 | 33.3 | 0
  Week 36: ACR 20 responders | 45.5 | 40.0 | 66.7 | 50.0
  Week 36: ACR 50 responders | 36.4 | 40.0 | 66.7 | 25.0
  Week 36: ACR 70 responders | 27.3 | 40.0 | 33.3 | 0
  Week 48: ACR 20 responders | 45.5 | 30.0 | 66.7 | 25.0
  Week 48: ACR 50 responders | 45.5 | 30.0 | 66.7 | 25.0
  Week 48: ACR 70 responders | 36.4 | 30.0 | 66.7 | 0
  Week 52: ACR 20 responders | 54.5 | 20.0 | 66.7 | 50.0
  Week 52: ACR 50 responders | 36.4 | 20.0 | 66.7 | 50.0
  Week 52: ACR 70 responders | 27.3 | 20.0 | 66.7 | 0

38. Secondary Outcome: Percent Change From Baseline in the Tender Joints Count and Swollen Joints Count at Weeks 4, 8, and 16
Description: Percent change from baseline in the tender joints and swollen joints counts at Weeks 4, 8, and 16 was evaluated.
Time Frame: Weeks 4, 8, and 16
Population: Population included randomized participants at Week 0 and who had a diagnosis of PsA at screening. Here 'n' (number analyzed) signifies the number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 10
percent change
  Week 4: Tender joints | -7.4 (22.22) | 41.1 (34.47) | -8.8 (117.56)
  Week 4: Swollen joints: number analyzed (Participants) | 8 | 10 | 6
  Week 4: Swollen joints | 14.1 (35.00) | 20.5 (39.50) | 22.2 (32.77)
  Week 8: Tender joints: number analyzed (Participants) | 9 | 10 | 9
  Week 8: Tender joints | -54.6 (188.70) | 47.3 (39.61) | 50.1 (58.06)
  Week 8: Swollen joints: number analyzed (Participants) | 8 | 10 | 6
  Week 8: Swollen joints | 29.5 (39.76) | 56.0 (42.33) | 50.0 (40.82)
  Week 16: Tender joints: number analyzed (Participants) | 9 | 10 | 9
  Week 16: Tender joints | -60.2 (86.58) | 47.0 (40.12) | 22.7 (126.76)
  Week 16: Swollen joints: number analyzed (Participants) | 8 | 10 | 6
  Week 16: Swollen joints | 22.7 (52.66) | 55.7 (46.71) | 79.2 (40.05)

39. Secondary Outcome: Percent Change From Baseline in the Tender Joints Count and Swollen Joints Count at Weeks 28, 36, 48, and 52
Description: Percent change from baseline in the tender joints and swollen joints counts at Weeks 28, 36, 48 and 52 was evaluated.
Time Frame: Weeks 28, 36, 48, and 52
Population: Population included participants who were randomized to Guselkumab at Week 0 or 16 and had a diagnosis of PsA at screening. Here 'n' signifies the number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 10 | 3 | 4
percent change
  Week 28: Tender joints: number analyzed (Participants) | 10 | 9 | 3 | 4
  Week 28: Tender joints | 54.9 (41.34) | 60.6 (46.80) | 33.3 (76.38) | -100.0 (81.65)
  Week 28: Swollen joint: number analyzed (Participants) | 10 | 6 | 3 | 3
  Week 28: Swollen joint | 66.0 (39.14) | 94.4 (8.61) | 66.1 (29.36) | 43.3 (60.28)
  Week 36: Tender joints: number analyzed (Participants) | 10 | 9 | 3 | 4
  Week 36: Tender joints | 69.7 (40.66) | 62.1 (47.33) | 33.3 (76.38) | 25.0 (95.74)
  Week 36: Swollen joint: number analyzed (Participants) | 10 | 6 | 3 | 3
  Week 36: Swollen joint | 55.2 (64.82) | 94.4 (13.61) | 84.7 (16.84) | 63.3 (32.15)
  Week 48: Tender joints: number analyzed (Participants) | 10 | 9 | 3 | 4
  Week 48: Tender joints | 53.9 (61.03) | 45.4 (73.14) | 50.0 (86.60) | 25.0 (95.74)
  Week 48: Swollen joint: number analyzed (Participants) | 10 | 6 | 3 | 3
  Week 48: Swollen joint | 72.4 (42.84) | 80.6 (34.02) | 82.8 (13.98) | 70.0 (26.46)
  Week 52: Tender joints: number analyzed (Participants) | 10 | 9 | 3 | 4
  Week 52: Tender joints | 67.8 (47.31) | 32.9 (72.40) | 66.7 (57.74) | 75.0 (50.00)
  Week 52: Swollen joint: number analyzed (Participants) | 10 | 6 | 3 | 3
  Week 52: Swollen joint | 84.5 (32.70) | 58.3 (55.53) | 88.9 (19.25) | 86.7 (23.09)

40. Secondary Outcome: Change From Baseline in the Tender Joints Count and Swollen Joints Count at Weeks 4, 8, and 16
Description: Change from baseline in the tender joints and swollen joints counts at Weeks 4, 8, and 16 was evaluated.
Time Frame: Baseline and Weeks 4, 8, 16
Population: Population included randomized participants at Week 0 and who had a diagnosis of PsA at screening.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 10
joints
  Week 4: Tender joints | 0.2 (0.63) | -3.8 (6.15) | -1.6 (4.74)
  Week 4: Swollen joints | -0.4 (0.97) | -1.2 (2.44) | -0.4 (1.58)
  Week 8: Tender joints | 0.9 (3.38) | -4.9 (9.24) | -2.6 (4.79)
  Week 8: Swollen joints | -1.9 (4.68) | -2.1 (2.55) | -2.2 (3.43)
  Week 16: Tender joints | 1.3 (2.06) | -3.9 (6.32) | -3.3 (5.17)
  Week 16: Swollen joints | -1.3 (3.56) | -2.3 (3.41) | -3.2 (4.37)

41. Secondary Outcome: Change From Baseline in the Tender Joints Count and Swollen Joints Count at Weeks 28, 36, 48, and 52
Description: Change from baseline in the tender joints and swollen joints counts at Weeks 28, 36, 48 and 52 was evaluated.
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 10 | 3 | 4
joints
  Week 28: Tender joints | -4.0 (6.03) | -4.1 (5.93) | -1.0 (2.00) | 1.8 (1.71)
  Week 28: Swollen joint | -2.5 (2.81) | -3.4 (4.35) | -9.7 (8.02) | -0.3 (0.96)
  Week 36: Tender joints | -3.8 (6.23) | -4.0 (5.08) | -1.0 (2.00) | -1.0 (2.16)
  Week 36: Swollen joint | -2.8 (3.46) | -3.6 (4.79) | -11.7 (8.62) | -1.0 (0.82)
  Week 48: Tender joints | -3.3 (7.18) | -3.0 (4.83) | -1.3 (2.08) | -1.0 (2.16)
  Week 48: Swollen joint | -2.9 (3.30) | -2.5 (3.87) | -11.7 (9.29) | -1.3 (1.26)
  Week 52: Tender joints | -7.0 (11.19) | -2.9 (4.58) | -1.7 (1.53) | -1.5 (1.73)
  Week 52: Swollen joint: number analyzed (Participants) | 10 | 6 | 3 | 3
  Week 52: Swollen joint | -3.2 (3.43) | -1.5 (4.09) | -12.7 (10.26) | -1.5 (1.29)

42. Secondary Outcome: Percent Change From Baseline in Patient's Assessment of Pain (VAS) at Weeks 4, 8, 16
Description: Percent change from baseline in Patient's Assessment of Pain (VAS) among participants who had a diagnosis of PsA at screening at Weeks 4, 8 and 16 was evaluated. Each participant assessed his/her pain associated with joint symptoms on each assessment day using a 100 mm VAS ranging from 0 millimeter (mm) (no pain) to 100 mm (the worst pain imaginable).
Time Frame: Baseline and Weeks 4, 8, 16
Population: Population included randomized participants at Week 0 and who had diagnosis of PsA at screening. Participants were analyzed according to assigned treatment they were randomized to, regardless of treatment they actually received. Here, N (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 7
percent change
  Week 4 | 13.70 (23.698) | 3.99 (78.918) | 10.32 (118.053)
  Week 8 | 2.36 (37.869) | 38.19 (43.951) | 45.15 (55.679)
  Week 16 | -0.73 (33.066) | 45.51 (34.419) | 62.11 (41.719)

43. Secondary Outcome: Percent Change From Baseline in Patient's Assessment of Pain (VAS) at Weeks 28, 36, 48, 52
Description: Percent change from baseline in Patient's Assessment of Pain (VAS) among participants who had a diagnosis of PsA at screening at Weeks 28, 36, 48 and 52 was evaluated. Each participant assessed his/her pain associated with joint symptoms on each assessment day using a 100 mm VAS ranging from 0 mm (no pain) to 100 mm (the worst pain imaginable).
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: Population included participants who were randomized to Guselkumab at Week 0 or 16 and had a diagnosis of PsA at screening. Here, N (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 7 | 3 | 4
Percent change
  Week 28 | -37.67 (339.724) | 73.28 (28.687) | 51.18 (30.418) | 40.96 (73.340)
  Week 36 | -26.65 (273.745) | 68.21 (40.538) | 71.92 (21.156) | 47.37 (46.079)
  Week 48 | 50.38 (74.874) | 57.65 (34.861) | 81.36 (12.019) | 74.08 (14.330)
  Week 52 | -30.54 (305.279) | 62.09 (40.678) | 77.06 (23.487) | 61.47 (67.467)

44. Secondary Outcome: Percent Change From Baseline in Patient's Global Assessment of Disease Activity at Weeks 4, 8, 16
Description: The participant's and physician's global assessments of disease activity were recorded on a VAS. The VAS for the participant's assessment ranges from "very well" (0 centimeter [cm]) to "very poor" (10 cm).
Time Frame: Baseline and Weeks 4, 8, 16
Population: Population included randomized participants at Week 0 and who had a diagnosis of PsA at screening. Here, N (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 6
percent change
  Week 4 | 12.55 (24.547) | 39.64 (38.514) | 58.81 (29.281)
  Week 8 | 2.50 (34.402) | 44.50 (39.328) | 63.10 (42.085)
  Week 16 | -6.52 (28.037) | 21.38 (71.545) | 75.70 (34.106)

45. Secondary Outcome: Percent Change From Baseline in Patient's Global Assessment of Disease Activity at Weeks 28, 36, 48, and 52
Description: The participant's and physician's global assessments of disease activity were recorded on a VAS. The VAS for the participant's assessment ranges from "very well" (0 cm) to "very poor" (10 cm).
Time Frame: Baseline and Weeks 28, 36, 48, 52
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 6 | 3 | 4
percent change
  Week 28 | -46.83 (346.499) | 71.26 (35.552) | 45.85 (35.019) | 61.23 (16.062)
  Week 36 | -48.87 (341.563) | 75.55 (33.992) | 51.95 (27.007) | 54.46 (27.386)
  Week 48 | 43.09 (109.254) | 58.36 (41.137) | 76.02 (24.470) | 67.60 (20.616)
  Week 52 | -20.17 (298.482) | 66.00 (36.151) | 71.59 (34.140) | 69.10 (47.796)

46. Secondary Outcome: Percentage of Participants Who Achieved Health Assessment Questionnaire-Disability Index (HAQ-DI) Response at Weeks 4, 8 and 16
Description: HAQ-DI response was defined as change of less than or equal to (<=) -0.3 from baseline in HAQ-DI score. HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area (that is, lower scores are indicative of better functioning).
Time Frame: Weeks 4, 8, and 16
Population: Population included randomized participants at Week 0 and who had a diagnosis of PsA at screening.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP)
Number analyzed (Participants) | 10 | 11 | 10
percentage of participants
  Week 4 | 10.0 | 36.4 | 10.0
  Week 8 | 20.0 | 45.5 | 20.0
  Week 16 | 0 | 54.5 | 30.0

47. Secondary Outcome: Percentage of Participants Who Achieved HAQ-DI Response at Weeks 28, 36, 48, 52
Description: as for outcome 46
Time Frame: Weeks 28, 36, 48, 52
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Number analyzed (Participants) | 11 | 10 | 3 | 4
percentage of participants
  Week 28 | 45.5 | 30.0 | 66.7 | 25.0
  Week 36 | 54.5 | 30.0 | 66.7 | 0
  Week 48 | 45.5 | 20.0 | 66.7 | 25.0
  Week 52 | 45.5 | 10.0 | 66.7 | 25.0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: The safety analysis set included all participants who received at least 1 study agent administration. In the safety analyses, participants were analyzed according to the treatment they actually received, regardless of the treatments they were randomized to.
Groups:
- Guselkumab 50 mg (CP): Participants stratified by the type of psoriasis (with or without PsA) received guselkumab 50 mg SC injection and placebo 100 mg at Week 0, Week 4, and Week 12.
- Guselkumab 100 mg (CP): Participants stratified by the type of psoriasis (with or without PsA) received guselkumab 100 mg SC injection and placebo 50 mg at Week 0, Week 4, and Week 12.
- Guselkumab 50 mg (After CP): Participants who completed CP continued to after CP period. At Week 16, participants in this group received placebo 50 mg and 100 mg to maintain blind. After Week 16, participants received guselkumab 50 mg and placebo 100 mg at Weeks 20, 28, 36, and 44.
- Guselkumab 100 mg (After CP): Participants who completed CP continued to after CP period. At Week 16, participants in this group received placebo 50 mg and 100 mg to maintain blind. After Week 16, participants received guselkumab 100 mg and placebo 50 mg at Weeks 20, 28, 36, and 44.
Arm/Group | Placebo (CP) | Guselkumab 50 mg (CP) | Guselkumab 100 mg (CP) | Guselkumab 50 mg (After CP) | Guselkumab 100 mg (After CP) | Placebo to Guselkumab 50 mg (After CP) | Placebo to Guselkumab 100 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 2/64 | 1/65 | 1/63 | 6/63 | 6/62 | 4/26 | 5/26
Other Adverse Events (participants affected / at risk) | 36/64 | 27/65 | 26/63 | 56/63 | 55/62 | 25/26 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=64) | Guselkumab 50 mg (CP) (N=65) | Guselkumab 100 mg (CP) (N=63) | Guselkumab 50 mg (After CP) (N=63) | Guselkumab 100 mg (After CP) (N=62) | Placebo to Guselkumab 50 mg (After CP) (N=26) | Placebo to Guselkumab 100 mg (After CP) (N=26)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macular Hole (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhegmatogenous Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial Prostatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gouty Tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to the Mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thalamus Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=64) | Guselkumab 50 mg (CP) (N=65) | Guselkumab 100 mg (CP) (N=63) | Guselkumab 50 mg (After CP) (N=63) | Guselkumab 100 mg (After CP) (N=62) | Placebo to Guselkumab 50 mg (After CP) (N=26) | Placebo to Guselkumab 100 mg (After CP) (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermoid Cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
External Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Corneal Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 4 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 3
Dental Caries (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 5 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 7 | 2 | 2 | 2
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Injection Site Discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 1 | 0 | 0 | 5 | 7 | 3 | 4
Injection Site Hypertrichosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Hypertrophy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Induration (General disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 1
Injection Site Pain (General disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 0 | 4 | 3 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 3
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 4 | 1 | 2
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 2
Hepatitis Alcoholic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2 | 5 | 0 | 6
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Diarrhoea Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 1 | 3 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Groin Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 2 | 0 | 1 | 3 | 0 | 0
Infectious Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 9 | 3 | 5 | 5
Lice Infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 14 | 8 | 38 | 31 | 14 | 14
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 5 | 5 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tinea Cruris (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 5 | 1 | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 2 | 2 | 4 | 1 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 5 | 1 | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Nerve Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 3 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Triglycerides Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Electrocardiogram Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Electrocardiogram QT Prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 1
Liver Function Test Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Weight Increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 6 | 0 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic Disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 9 | 6 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 7 | 6 | 2 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Blepharal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 6 | 2 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radial Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 2 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasal Mucosal Erosion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0
Pharyngeal Paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5 | 1 | 0 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 4 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 7 | 3 | 5
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 0
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 2
Palmoplantar Pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 3 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 11 | 0 | 0 | 0 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 4 | 1 | 3
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0 | 7 | 6 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.